CLINICAL TRIAL: NCT03549351
Title: Prospective Evaluation of Measurable Residual Disease in Intensively Treated Patients With Acute Myeloid Leukemia (AML) as Surrogate Endpoint for Survival
Brief Title: Evaluation of Measurable Residual Disease in Patients With Acute Myeloid Leukemia as Surrogate Endpoint for Survival
Acronym: PERDAM
Status: Terminated | Type: Observational
Why Stopped: Study turned out no longer feasible
Sponsor: University Hospital Heidelberg (Other)
Collaborators: University Hospital Dresden (Other); German Cancer Research Center (Other)
Responsible Party: Principal Investigator, Prof. Dr. Richard F Schlenk, Head of NCT trials center, University Hospital Heidelberg
Other Study IDs: NCT-2018-0554
Record Dates: First submitted 2018-05-07; First posted 2018-06-08 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Leukemia, Myeloid, Acute; measurable residual disease; surrogate endpoint; multiparameter flow cytometry
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood Samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measurable residual disease measured by flow cytometry — Measurable residual disease measured by flow cytometry

SUMMARY:
Objectives To demonstrate that measurable residual disease assessed by multiparameter flow cytometry during intensive treatment is a surrogate for overall survival and thus an early read-out for drug efficacy Study design Surrogate endpoint trial to establish that measurable residual disease assessed by multiparameter flow cytometry during intensive treatment is a surrogate for overall survival

DETAILED DESCRIPTION:
Acute myeloid leukemia is a genetically and phenotypically heterogeneous disorder with an incidence of 3 to 4 per 100 000 men and women per year and a median age at diagnosis of about 70 years. Prognosis, especially in older patients, has remained very poor. In patients considered suitable for intensive chemotherapy, the combination of an anthracycline and cytarabine remains the standard of care. For patients achieving a complete remission (CR), postremission therapy (PRT) ranging from chemotherapy to allogeneic hematopoietic stem cell transplantation is required; intensive PRT is still under debate in older patients. Beyond pre-treatment genetics-based risk stratification, measurable residual disease (MRD) during treatment and follow up emerges as an important prognostic factor in first CR. Furthermore, MRD may provide a tool for a read-out of therapeutic efficacy. In this diagnostic meta-study the investigators intend to measure MRD using multiparameter flow cytometry across up-front randomized clinical trials which in total will accrue more than 1000 patients. According to the leukemia-associated phenotype at diagnosis or the different-from-normal approach, MRD will be assessed early (after induction) and late (after consolidation) during treatment. The aim of the study is to show that levels of MRD measured early during treatment are closely related to overall survival and thus may serve as an early surrogate. There is a growing public demand that new, promising drugs are approved for therapy as rapidly as possible. Therefore, it is of great interest to obtain these approvals based on early biomarker endpoints such as MRD rather than on long-term survival endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia according to the WHO classification
* Informed consent in place for a randomized study of the Study Alliance Leukemia (SAL) including the Heidelberg Leukemia Network (HeLeNe) covering assessment of MRD by MPFC in the reference laboratories in Heidelberg and Dresden.

Exclusion Criteria:

* No signed informed consent compliant with the requirements of PERDAM

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with AML participating in interventional prospective randomized trials of the Study Alliance Leukemia (SAL) including the Heidelberg Leukemia Network (HeLeNe)
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2022-09-11 (Actual)

PRIMARY OUTCOMES:
Correlation between Measurable Residual Disease (MRD) and Survival with respect to treatment effects | after 3 and 6 years
  MRD will be assessed using multiparameter flow cytometry early (after induction / salvage).
  Survival will be assessed continuously. After 3 and 6 years correlation between MRD and survival will be analysed with respect to treatment effects to assess if MRD may serve as surrogate endpoint.
  If levels of MRD measured early during treatment are closely related to overall survival and thus may serve as an early surrogate will be assessed yearly.

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Schlenk, Prof. Dr., Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT03549351/Prot_SAP_000.pdf